CLINICAL TRIAL: NCT00754494
Title: A Phase IIa Randomized, Double-Blind Trial of Erlotinib in Inhibiting EGF Receptor Signaling in Aberrant Crypt Foci of the Colon
Brief Title: Erlotinib Hydrochloride in Treating Patients With Stage I-III Colorectal Cancer or Adenoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NCI-2012-02984; UCI06-8-01; N01CN35160 (NIH); CDR0000614277 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Results first posted 2015-01-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2014-03

CONDITIONS: Adenomatous Polyp; Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage I Colon Cancer; Stage I Rectal Cancer; Stage IIA Colon Cancer; Stage IIA Rectal Cancer; Stage IIB Colon Cancer; Stage IIB Rectal Cancer; Stage IIC Colon Cancer; Stage IIC Rectal Cancer; Stage IIIA Colon Cancer; Stage IIIA Rectal Cancer; Stage IIIB Colon Cancer; Stage IIIB Rectal Cancer; Stage IIIC Colon Cancer; Stage IIIC Rectal Cancer
MeSH Terms: conditions — Adenomatous Polyps; Colonic Neoplasms; Rectal Neoplasms | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- Erlotinib Hydrochloride (25 mg) (Experimental): Patients receive 25mg of erlotinib hydrochloride PO and one 100 mg of placebo and one 25 mg of placebo PO QD.
  Interventions: Drug: erlotinib hydrochloride; Other: placebo; Other: laboratory biomarker analysis
- Erlotinib Hydrochloride (50 mg) (Experimental): Patients receive 50 mg of erlotinib hydrochloride PO and one 100 mg of placebo PO QD.
  Interventions: Drug: erlotinib hydrochloride; Other: placebo; Other: laboratory biomarker analysis
- Erlotinib Hydrochloride (100 mg) (Experimental): Patients receive 100 mg of erlotinib hydrochloride PO and two 25 mg of placebo PO QD.
  Interventions: Drug: erlotinib hydrochloride; Other: placebo; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given PO
  Other Names: CP-358,774; erlotinib; OSI-774
Other: placebo — Given PO
  Other Names: PLCB
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II trial is studying how well erlotinib hydrochloride works in treating patients with stage I-III colorectal cancer or adenoma. Erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Erlotinib hydrochloride may also stop tumors from growing or coming back

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test the hypothesis that erlotinib (erlotinib hydrochloride) doses as low as 25 mg will decrease aberrant crypt foci (ACF) phosphorylated extracellular signal-regulated kinases (pERK) levels from baseline (pre) to post erlotinib treatment.

SECONDARY OBJECTIVES:

I. To test the hypothesis that additional epidermal growth factor (EGF) inducible biomarkers will decrease from baseline (pre) to post treatment with erlotinib 25 mg, 50 mg or 100 mg orally (PO) once daily (QD) therapy.

II. To determine the mean decrease from baseline of the ACF: normal mucosa pERK ratio pre and post 8-30 days of erlotinib.

III. To determine erlotinib concentration in plasma and colorectal tissue at 25 mg, 50 mg and 100 mg doses after 8-30 days of therapy.

IV. To determine the incidence of rash, diarrhea and other side effects of low dose erlotinib.

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

ARM I: Patients receive 100 mg of erlotinib hydrochloride PO and two 25 mg of placebo PO QD.

ARM II: Patients receive 50 mg of erlotinib hydrochloride PO and one 100 mg of placebo PO QD.

ARM III: Patients receive 25 mg of erlotinib hydrochloride PO and one 100 mg of placebo and one 25 mg of placebo PO QD.

In all arms, treatment continues for 8-30 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 to 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants with one or more of the following criteria will be eligible to participate:

  * History of Stage I-III colorectal cancer, not treated in the past 6 months with no anticipated treatment in the next 3 months
  * Adenoma ≥ 1 cm in size
  * 3 or more adenomas (of any size) removed at one colonoscopy within past 6 years
  * Sessile serrated adenoma ≥ 5 mm in size
  * Adenoma (of any size) with villous features (villous, tubulovillous)
  * Adenoma (of any size) with high grade dysplasia
* Participants are eligible for randomization into the treatment phase of the trial if they are found to have ≥ 4 ACFs at either baseline colonoscopy or baseline flexible sigmoidoscopy
* Blood tests at screening which meet the following criteria:
* WBC > 3000/mm^3
* Platelets > 100,000/mm^3
* Hemoglobin > 10g/dl
* Plasma creatinine of < 1.6mg/dl
* Total bilirubin < 1.5 x the upper limit of normal
* Serum ALT < 1.5 x the upper limit of normal
* Serum AST < 1.5 x the upper limit of normal
* ECOG performance status 0-1
* Women of child-bearing potential and men taking study drug must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* Ability to understand, as well as sign the written informed consent document
* If a woman is of child-bearing potential, she must have a negative pregnancy test prior to study entry; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately

Exclusion Criteria:

* History of Inflammatory Bowel Disease (IBD)
* History of interstitial lung disease or chronic lung disease
* Smoking within the past 3 months
* Increased bleeding risk from rectal biopsy (Patients receiving aspirin or plavix can be enrolled)
* Patients receiving warfarin or coumadin
* Uncontrollable diarrhea of any cause
* Patients, including rectal cancer patients, that have received prior radiation to the rectum or pelvis
* Participants taking a known significant CYP 3A4 inducer or inhibitor; known significant inducers/inhibitors include: amprenavir, aprepitant, atazanavir, carbamazepine, clarithromycin, conivaptan, diltiazem, darunavir/ritonavir, dronedarone, erythromycin, fluconazole, fosamprenavir, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, phenytoin, posaconazole, rifampin, ritonavir, St. John's wort, saquinavir, telithromycin, tipranavir/ritonavir, verapamil, voriconazole
* Women who are pregnant or breast-feeding
* Active keratoconjunctivitis, or corneal surgery in the past three weeks
* Any medical or psychosocial condition that could jeopardize the subject's participation in and compliance to the study
* Participants who are taking any other investigational pharmaceutical agents
* Previous history of sensitivity to erlotinib, Iressa, or Erbitux, such as a rash that is uncontrollable by topical steroids and/or antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-07; Primary Completion 2012-10 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Morgan, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (3):
- United States (3):
  - VA Long Beach Healthcare System, Long Beach, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of Illinois at Chicago, Chicago, Illinois

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (25 mg): Patients receive 25mg of erlotinib hydrochloride PO and one 100 mg of placebo and one 25 mg of placebo PO QD.
  erlotinib hydrochloride: Given PO
  placebo: Given PO
  laboratory biomarker analysis: Correlative studies
- Arm II (50 mg): Patients receive 50 mg of erlotinib hydrochloride PO and one 100 mg of placebo PO QD.
  erlotinib hydrochloride: Given PO
  placebo: Given PO
  laboratory biomarker analysis: Correlative studies
- Arm III (100 mg): Patients receive 100 mg of erlotinib hydrochloride PO and two 25 mg of placebo PO QD.
  erlotinib hydrochloride: Given PO
  placebo: Given PO
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Arm I (25 mg) | Arm II (50 mg) | Arm III (100 mg)
Started | 15 | 15 | 15
Completed | 13 | 15 | 14
Not Completed | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (25 mg) | Arm II (50 mg) | Arm III (100 mg) | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.67 (4.43) | 62.47 (6.03) | 60.67 (7.42) | 62.27 (6.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 5 | 8
  Male | 13 | 14 | 10 | 37

OUTCOME MEASURES:

1. Primary Outcome: Change in ACF pERK Levels
Description: Quantification will be performed by Western blot analysis. Tested using paired t-test with a two-sided significance level of 0.05.
Time Frame: From baseline to post-treatment (up to 30 days)
Population: Change in ACF pERK levels not reported as the assay did not demonstrate signaling
Groups:
- Arm I (25 mg): Patients receive 25mg of erlotinib hydrochloride PO and one 100 mg of placebo and one 25 mg of placebo PO QD.
  erlotinib hydrochloride: Given PO
  placebo: Given PO
  laboratory biomarker analysis: Correlative studies
  The range of days on treatment is 10 to 29 days
- Arm II (50 mg): Patients receive 50 mg of erlotinib hydrochloride PO and one 100 mg of placebo PO QD.
  erlotinib hydrochloride: Given PO
  placebo: Given PO
  laboratory biomarker analysis: Correlative studies
  The range of days on treatment is 8 to 28 days
- Arm III (100 mg): Patients receive 100 mg of erlotinib hydrochloride PO and two 25 mg of placebo PO QD.
  erlotinib hydrochloride: Given PO
  placebo: Given PO
  laboratory biomarker analysis: Correlative studies
  The range of days on treatment is 7 to 23 days
Arm/Group | Arm I (25 mg) | Arm II (50 mg) | Arm III (100 mg)
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Change in EGF-inducible Markers - pEGFR in Normal Mucosa
Description: pEGFR expression levels were quantified by immunoblotting and calculated as the ratio of the pEGFR signals to reference signals. A log-transformation of pEGFR was utilized in primary analyses. The general linear model was used to estimate and compare the relative change in median pEGFR with adjustment for actin as a normalizing factor. The estimated relative change (post:pre) in the median, corresponding 95% confidence interval, and p-value for testing the null hypothesis of equal medians comparing pre- and post-measurements were reported.
Time Frame: From baseline to post-treatment (up to 30 days)
Population: Outcome measure data is reported based on the evaluable samples collected and available results.
Measure: Geometric Mean (95% Confidence Interval); unit: expression level
Arm/Group | Arm I (25 mg) | Arm II (50 mg) | Arm III (100 mg)
Number analyzed (Participants) | 14 | 14 | 13
expression level | 0.84 [0.27 to 2.58] | 1.65 [0.87 to 3.10] | 0.97 [0.68 to 1.38]
Statistical Analysis 1: Comparison: Arm I (25 mg); A log-transformation of pEGFR was utilized in primary analyses because of the highly skewed distribution observed in this outcome. The general linear model was used to estimate and compare the relative change in median pEGFR with adjustment for actin as a normalizing factor. The estimated relative change (post:pre) in the median, corresponding 95% confidence interval, and p-value for testing the null hypothesis of equal medians comparing pre- and post-measurements were reported; Test type: Superiority or Other; p = 0.762, General Linear Model
Statistical Analysis 2: Comparison: Arm II (50 mg); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.125, General Linear Model
Statistical Analysis 3: Comparison: Arm III (100 mg); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.855, General Linear Model

3. Secondary Outcome: Change in EGF-inducible Markers - Total EGFR in Normal Mucosa
Description: Total EGFR expression levels were quantified by immunoblotting and calculated as the ratio of the total EGFR signals to reference signals. A log-transformation of total EGFR was utilized in primary analyses. The general linear model was used to estimate and compare the relative change in median total EGFR with adjustment for actin as a normalizing factor. The estimated relative change (post:pre) in the median, corresponding 95% confidence interval, and p-value for testing the null hypothesis of equal medians comparing pre- and post-measurements were reported.
Time Frame: From baseline to post-treatment (up to 30 days)
Population: Outcome measure data is reported based on the evaluable samples collected and available results.
Measure: Geometric Mean (95% Confidence Interval); unit: expression level
Arm/Group | Arm I (25 mg) | Arm II (50 mg) | Arm III (100 mg)
Number analyzed (Participants) | 14 | 14 | 13
expression level | 2.02 [0.44 to 9.40] | 1.91 [0.91 to 4.00] | 1.23 [0.88 to 1.72]
Statistical Analysis 1: Comparison: Arm I (25 mg); A log-transformation of total EGFR was utilized in primary analyses because of the highly skewed distribution observed in this outcome. The general linear model was used to estimate and compare the relative change in median total EGFR with adjustment for actin as a normalizing factor. The estimated relative change (post:pre) in the median, corresponding 95% confidence interval, and p-value for testing the null hypothesis of equal medians comparing pre- and post-measurements were reported; Test type: Superiority or Other; p = 0.369, General Linear Model
Statistical Analysis 2: Comparison: Arm II (50 mg); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.085, General Linear Model
Statistical Analysis 3: Comparison: Arm III (100 mg); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.233, General Linear Model

4. Secondary Outcome: Change in EGF-inducible Markers - pEGFR in ACF
Description: pEGFR expression levels were quantified by immunoblotting and calculated as the ratio of the pEGFR signals to reference signals. A log-transformation of pEGFR was utilized in primary analyses. The general linear model was used to estimate and compare the relative change in median total EGFR with adjustment for actin as a normalizing factor. The estimated relative change (post:pre) in the median, corresponding 95% confidence interval, and p-value for testing the null hypothesis of equal medians comparing pre- and post-measurements were reported.
Time Frame: From baseline to post-treatment (up to 30 days)
Population: Outcome measure data is reported based on the evaluable samples collected and available results.
Measure: Geometric Mean (95% Confidence Interval); unit: expression level
Arm/Group | Arm I (25 mg) | Arm II (50 mg) | Arm III (100 mg)
Number analyzed (Participants) | 14 | 14 | 14
expression level | 1.19 [0.57 to 2.48] | 1.93 [1.07 to 3.48] | 1.40 [0.78 to 2.53]
Statistical Analysis 1: Comparison: Arm I (25 mg); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.651, General Linear Model
Statistical Analysis 2: Comparison: Arm II (50 mg); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.030, General Linear Model
Statistical Analysis 3: Comparison: Arm III (100 mg); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.261, General Linear Model

5. Secondary Outcome: Change in EGF-inducible Markers - Total EGFR in ACF
Description: as for outcome 3
Time Frame: From baseline to post-treatment (up to 30 days)
Population: Outcome measure data is reported based on the evaluable samples collected and available results.
Measure: Geometric Mean (95% Confidence Interval); unit: expression level
Arm/Group | Arm I (25 mg) | Arm II (50 mg) | Arm III (100 mg)
Number analyzed (Participants) | 14 | 14 | 14
expression level | 1.33 [0.38 to 4.61] | 2.22 [1.08 to 4.54] | 1.94 [0.92 to 4.09]
Statistical Analysis 1: Comparison: Arm I (25 mg); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.654, General Linear Model
Statistical Analysis 2: Comparison: Arm II (50 mg); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.030, General Linear Model
Statistical Analysis 3: Comparison: Arm III (100 mg); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.083, General Linear Model

6. Secondary Outcome: ACF: Normal Mucosa pERK Ratio
Description: Quantification will be performed by Western blot analysis. Tested using analysis of variance with subsequent pairwise comparisons using the Tukey method to adjust for multiple comparisons.
Time Frame: Up to day 30
Population: ACF: pERK ratio not reported as the assay did not demonstrate signaling in ACF pERK levels
Arm/Group | Arm I (25 mg) | Arm II (50 mg) | Arm III (100 mg)
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Plasma Erlotinib Concentration (ng/mL)
Description: Will be quantified in biopsy samples using appropriate descriptive statistics (means and standard deviations).
Time Frame: Up to day 30
Population: Outcome measure data is reported based on the evaluable samples collected and available results.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm I (25 mg) | Arm II (50 mg) | Arm III (100 mg)
Number analyzed (Participants) | 14 | 14 | 13
ng/mL | 232.29 (160.6) | 486.56 (211.8) | 1280.84 (788.3)

8. Secondary Outcome: Plasma OSI-420 Concentration (ng/mL)
Description: Will be quantified in biopsy samples using appropriate descriptive statistics (means and standard deviations).
Time Frame: Up to day 30
Population: Outcome measure data is reported based on the evaluable samples collected and available results.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm I (25 mg) | Arm II (50 mg) | Arm III (100 mg)
Number analyzed (Participants) | 13 | 14 | 13
ng/mL | 17.77 (12.3) | 33.87 (14.1) | 117.98 (84.5)

9. Secondary Outcome: Normal Mucosa Erlotinib Concentration (ng/mg)
Description: Will be quantified in biopsy samples using appropriate descriptive statistics (means and standard deviations).
Time Frame: Up to day 30
Population: Outcome measure data is reported based on the evaluable samples collected and available results.
Measure: Mean (Standard Deviation); unit: ng/mg
Arm/Group | Arm I (25 mg) | Arm II (50 mg) | Arm III (100 mg)
Number analyzed (Participants) | 12 | 12 | 12
ng/mg | 0.36 (0.18) | 1.38 (1.23) | 3.25 (4.62)

10. Secondary Outcome: Normal Mucosa OSI-420 Concentration (ng/mg)
Description: Will be quantified in biopsy samples using appropriate descriptive statistics (means and standard deviations).
Time Frame: Up to day 30
Population: Outcome measure data is reported based on the evaluable samples collected and available results.
Measure: Mean (Standard Deviation); unit: ng/mg
Arm/Group | Arm I (25 mg) | Arm II (50 mg) | Arm III (100 mg)
Number analyzed (Participants) | 4 | 10 | 11
ng/mg | 0.04 (0.01) | 0.17 (0.15) | 0.29 (0.24)

11. Secondary Outcome: Number of Participants Reported at Least 1 Side Effect During the Study
Description: Described for each arm using frequencies. The onset of adverse events is between randomization date and off-study date.
Time Frame: Up to 9 weeks
Measure: Number; unit: participants
Arm/Group | Arm I (25 mg) | Arm II (50 mg) | Arm III (100 mg)
Number analyzed (Participants) | 15 | 15 | 15
participants
  At least 1 adverse event reported | 12 | 13 | 13
  No adverse event reported | 3 | 2 | 2

12. Secondary Outcome: Number of Participants Reported at Least 1 Rash Side Effect During the Study
Description: Described for each arm using frequencies.
Time Frame: Up to 9 weeks
Measure: Number; unit: participants
Arm/Group | Arm I (25 mg) | Arm II (50 mg) | Arm III (100 mg)
Number analyzed (Participants) | 15 | 15 | 15
participants
  At least 1 rash AE reported | 5 | 6 | 12
  No rash AE reported | 10 | 9 | 3

13. Secondary Outcome: Number of Participants Reported at Least 1 Diarrhea Side Effect During the Study
Description: Described for each arm using frequencies.
Time Frame: Up to 9 weeks
Measure: Number; unit: participants
Arm/Group | Arm I (25 mg) | Arm II (50 mg) | Arm III (100 mg)
Number analyzed (Participants) | 15 | 15 | 15
participants
  At least 1 diarrhea AE reported | 4 | 4 | 5
  No diarrhea AE reported | 11 | 11 | 10

ADVERSE EVENTS:
Time Frame: The onset date of adverse event is between the randomization date and the date of off-study, up to 95 days.
Arm/Group | Arm I (25 mg) | Arm II (50 mg) | Arm III (100 mg)
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 12/15 | 13/15 | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (25 mg) (N=15) | Arm II (50 mg) (N=15) | Arm III (100 mg) (N=15)
CHEST PAIN (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (25 mg) (N=15) | Arm II (50 mg) (N=15) | Arm III (100 mg) (N=15)
80% DIMINISHED SEBORRHEIC KERATOSIS SKIN LESIONS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
ALLERGIC REACTION: RASH ON THE FACE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
BLOODY NOSE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
BLUE COLORED URINE (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
BLUE/GREEN COLORED URINE (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
BLURRING OF VISION (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
CANKER SORES (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
CLEARED UP ACNE ON MY FOREHEAD (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
COLD (General disorders) | 1 (1) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
DEEP BRUISED LFT LEG PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 3 (3) | 3 (4) | 4 (5)
DIARRHEA-FREQUENT BM'S (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
DRY & ITCHY SKIN (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
DRY EYE (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
DRY EYES (Eye disorders) | 0 (0) | 2 (2) | 1 (1)
DRY ITCHY EYE (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 5 (5)
DRY SKIN AROUND NOSE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
DRY SKIN ON NOSE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
DRY SKIN-(LEGS) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
DRYNESS OF EYES (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
DRYNESS OF SKIN ON FACE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
DULL SORENESS IN LEG (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
EARACHE (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
FACE PIMPLES (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
FACE SORE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 0 (0) | 3 (3)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
FLU (General disorders) | 0 (0) | 1 (1) | 0 (0)
FOLLICULAR RASH ON TORSO (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
HEARTBURN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
INCARCERATED HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
IRRITABLE-MOOD ALTERATION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
ITCHINESS OF EYES (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
LIGHT HEADED (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
LOOSE STOOLS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
LOSS OF APPETITE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
LOTS OF GAS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
MILD DIARRHEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
MILD INDIGESTION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
MILD RASH IN THE BUTTOCK (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
MOUTH SORES (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
NOSE BLEED (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PAIN ON ABDOMEN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
PAIN ON FOOT (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
PAINFUL ITCHY & TENDER SCALP (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 4 (4)
RASH ON CHEST (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
RASH ON FACE, CHEST AND SHOULDER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
RASH ON FACE, CHEST, AND BEHIND EARS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
RASH ON FACE, SCALP AND CHEST (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
RASH ON FACE, SCALP, CHEST (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
RASH ON FACE, SCALP, CHEST, BACK, EXTREMITIES (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
RASH ON FOOT (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
RASH ON FOREHEAD/NOSE/CHEST (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
RAW NOSE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
RED ITCHY FACE RASH ON CHEEKS & NOSE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
RED PUFFY EYES (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
RED RASH-FACE PEELING & NOW WHITE HEAD PIMPLES (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
RED RASH-FACE,NOSE, & CHEST (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
RED RASH-FACE-NECK-CHEST & SCALP-ITCHY (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
RED,BUMPY FACE & CHEST RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
RUNNY NOSE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
SEEING BLACK SPOTS AND FLASHING LIGHTS IN LEFT EYE (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
SHORT OF BREATH EASILY (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
SHORT OF BREATH-DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
SWOLLEN FACE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
SWOLLEN LEFT KNEE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
ULCER ON MUCOUS MEMBRANE IN MOUTH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
VOMIT (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less